CLINICAL TRIAL: NCT05639959
Title: Efficacy and Safety of New Mometasone Furoate Nasal Spray Formulation in Acute Rhinosinusitis Patients: A Randomized Clinical Trial
Status: Completed | Type: Observational
Sponsor: Saffron Pharma (Industry)
Responsible Party: Principal Investigator, Yasir Mehmood Mehmood, Dr Yasir Mehmood, Saffron Pharma
Other Study IDs: QA/CT/001
Record Dates: First submitted 2022-11-27; First posted 2022-12-07 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-11

CONDITIONS: Acute Rhinosinusitis
MeSH Terms: interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Commercial product group: group who are taking commercial nasal spray products
  Interventions: Drug: Mometasone Nasal 50 Mcg/Inh Nasal Spray; Device: Nasal spray
- New formulation product group: who are taking new formulation nasal spray product with same strength
  Interventions: Drug: Mometasone Nasal 50 Mcg/Inh Nasal Spray; Device: Nasal spray

INTERVENTIONS:
Drug: Mometasone Nasal 50 Mcg/Inh Nasal Spray — Mometasone furoate nasal spray effectively reduced total and individual symptoms scores in patients with allergic rhinitis.
  Other Names: Hivate
Device: Nasal spray — device can work properly for actuation during trials

SUMMARY:
Seasonal and perennial allergic rhinitis, acute rhino sinusitis, and nasal polyposis are examples of common inflammatory disorders of the airway that significantly reduce patient health and quality of life. Intranasal corticosteroids are advised as part of treatment plans for each of these illnesses since they help to reduce inflammation and thus symptoms.

Objective In order to assess the effectiveness and safety of a new nano formulation of Mometasone furoate nano-nasal spray (FM-NNS) for the treatment of allergic rhinitis. Mometasone Furoate Nano-nasal spray (FM-NNS) was compared with commercial available nasal spray named as MFNS.

DETAILED DESCRIPTION:
Background Seasonal and perennial allergic rhinitis, acute rhino sinusitis, and nasal polyposis are examples of common inflammatory disorders of the airway that significantly reduce patient health and quality of life. Intranasal corticosteroids are advised as part of treatment plans for each of these illnesses since they help to reduce inflammation and thus symptoms.

Objective In order to assess the effectiveness and safety of a new nano formulation of Mometasone furoate nano-nasal spray (FM-NNS) for the treatment of allergic rhinitis. Mometasone Furoate Nano-nasal spray (FM-NNS) was compared with commercial available nasal spray named as MFNS.

ELIGIBILITY:
Inclusion Criteria:

1. Children and adults of age (10-50) who had a diagnosis of rhinitis
2. Ability and willingness to understand and provide informed consent.

Exclusion Criteria:

1. Known current pregnancy.
2. Current hospitalization.
3. Unable to complete online questionnaires or adhere to study requirements.
4. Kidney failure or dialysis; severe liver disease or cirrhosis.
5. Any parathyroid conditions.
6. Known current pregnancy.
7. History of SARS-CoV-2 infection.

Ages: 10 Years to 50 Years | Sex: All
Age Groups: Child, Adult
Study Population: Ages Eligible for Study: 10 Years to 50 Years older Sexes Eligible for Study: All Accepts Healthy Volunteers: No Children and adults of any age who had a diagnosis of rhinitis sicca, symptoms of dry nose brought on by the use of specific drugs, or who were receiving concurrent treatment for allergies or rhinosinusitis were eligible for the study
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-09-10 (Actual); Primary Completion 2022-11-06 (Actual); Study Completion 2022-11-06 (Actual)

PRIMARY OUTCOMES:
congestion | 3 weeks
  The primary end outcomes were change from baseline in the subject's congestion and/or blockage score averaged throughout the first month of treatment and change from baseline in the physician's assessment of Allergic rhinitis.

CONTACTS AND LOCATIONS:
Locations (1):
- Saffron Pharmaceutical, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No